CLINICAL TRIAL: NCT03988205
Title: The Feasibility of Safely Managing Patients Receiving Induction With Liposomal Daunorubicin and Cytarabine (CPX-351) for Acute Myeloid Leukemia (AML) in an Outpatient Environment
Brief Title: Patients Receiving Induction With Liposomal Daunorubicin and Cytarabine (CPX-351) for Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Laura Michaelis, Associate Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO34597
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Results first posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Acute Myeloid Leukemia; Outpatient; CPX-351; Vyxeos®; Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — CPX-351; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): The study intervention is the application of a prescribed outpatient care model including a nurse teacher educational program and quality of life surveys for both subjects and caregivers. Induction therapy and medical follow up are performed without prophylactic admission to an inpatient facility. Subjects will also receive CPX-351 according to FDA approval, to subjects who meet medical and logistical criteria for study enrollment.
  Interventions: Behavioral: Outpatient Care Model; Drug: CPX-351

INTERVENTIONS:
Behavioral: Outpatient Care Model — Outpatient care model includes a nurse teacher educational program, scheduled outpatient visit protocol, and quality of life surveys for both subjects and caregivers.
Drug: CPX-351 — CPX-351 is administered, according to FDA approval, to subjects who meet medical and logistical criteria for study enrollment.
  Other Names: Cytarabine; Vyxeos®

SUMMARY:
This is a single-arm, single-site run-in phase (six subjects) followed by a multicenter continuation phase (114 subjects), Phase IV study. Eligible subjects will be receiving CPX-351 as their usual medical care administered according to FDA approval, as a condition for participation.

DETAILED DESCRIPTION:
This is an open-label, non-randomized study of a non-drug intervention in subjects receiving CPX-351 as their usual medical care administered according to its FDA approval. The study intervention is the application of a prescribed outpatient care model, including a nurse teacher educational program and quality of life surveys for both subjects and caregivers, in subjects who meet medical and logistical criteria. Induction therapy and medical follow-up are performed without prophylactic admission to an inpatient facility.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with newly diagnosed acute myeloid leukemia who are eligible for treatment with CPX-351 therapy according to the FDA approval and indication: therapy-related AML (t-AML) or AML with myelodysplasia-related changes (AML-MRC).
2. Age ≥ 18 years
3. Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1 (or Karnofsky Performance Status equivalent of 70 or above).
4. Total bilirubin ≤ 3 mg/dL.
5. Creatinine clearance > 30 mL/min by Cockcroft/Gault equation.
6. Adequate cardiac function, as assessed by ejection fraction( ≥50% for anthracycline therapy) via multiple-gated acquisition (MUGA) or echocardiogram.
7. Total white blood cell count of ≤ 20,000/µL on peripheral blood assessment (hydrea and/or leukapheresis allowed).
8. No evidence of active, uncontrolled infection.
9. No evidence of clinically significant disseminated intervascular coagulation (DIC)
10. No clinically significant abnormalities in core vital signs like heart rate, blood pressure or oxygenation which require inpatient evaluation or monitoring.
11. In the opinion of the enrolling physician, the subject is not at risk for clinically significant tumor lysis syndrome based on clinical assessment, complete blood count (CBC), comprehensive metabolic panel (CMP), uric acid, and lactate dehydrogenase (LDH).
12. In the opinion of the enrolling physician, no medical conditions that preclude the subject or the primary caregiver from transportation to and from the outpatient clinical care facility.
13. Both subject and the identified primary caregiver(s) signed informed consent.
14. In the opinion of the enrolling physician, there are no medical contraindications to outpatient induction and management.
15. Male subjects, even if surgically sterilized (i.e., status post vasectomy), must agree to one of the followings:

    * Practice effective barrier contraception during the entire study period and through six months after the last dose of CPX-351, OR
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)

Female subjects must meet one of the followings:

* Postmenopausal for at least one year before enrollment, OR
* Surgically sterile (i.e., undergone a hysterectomy or bilateral oophorectomy), OR
* If the subject is of childbearing potential (defined as not satisfying either of the above two criteria), she must agree to practice two acceptable methods of contraception (combination methods require use of two of the following: diaphragm with spermicide, cervical cap with spermicide, contraceptive sponge, male or female condom, hormonal contraceptive) from the time of signing of the informed consent form through six months after the last dose of CPX-351, OR o Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable contraception methods.)

Logistical Inclusion Criteria

1. The subject must be able to reside within approximately 45 minutes of the hospital where induction therapy is administered, during normal driving conditions (in the opinion of the enrolling physician), until count recovery or 60 days post-treatment, whichever comes first
2. The enrolling physician must verify and attest that the subject has a primary caregiver meeting all the following criteria:

   * Reside with the subject.
   * Be able to care for the subject full time or arrange to share full-time care with secondary caregivers.
   * Provide transportation.
   * Respond to clinical issues that arise.
   * Communicate with subject and physician in a timely manner.
3. The nurse teacher must verify that the subject and primary caregiver have completed and adequately understand the study-dictated nurse teacher educational program.
4. The nurse teacher must verify the subject and primary caregiver have capacity to comply with outpatient management program.
5. The subject must have reliable, working telephone access.
6. The subject must be willing and able to attend all protocol-dictated visits and be seen frequently as an outpatient at the clinical care facility where induction therapy is administered.

Exclusion Criteria:

1. Pregnant women (per pregnancy test in women of childbearing potential) or women who are breast-feeding.
2. Subjects currently receiving any investigational agents.
3. Subjects must not have current evidence of another malignancy that requires treatment.
4. Subjects diagnosed with Wilson's disease and/or copper-related metabolic disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Michaelis, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.34 (.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Adherent to Recommendations
Description: This measure will record the number subjects who adhere to outpatient follow-up appointments and readmission recommendations. Subjects completing 95% of their recommended outpatient visits will be considered to be adherent to the recommendations.
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 3
Participants | 3

2. Primary Outcome: Number of Participants Adherent to Readmission Recommendations
Description: This measure will record the number of subjects who complete as 100% compliance with medical provider recommendations to be admitted to the hospital (except for reasons of adopting a palliative or hospice approach to care). Subjects not achieving a 100% rate of compliance will be considered non-adherent to the recommendations.
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Fever (General disorders) | 1 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (11)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Blood bicarbonate decreased (Investigations) | 1 (3)
Investigations - Other, specify (Investigations) | 1 (15)
Lymphocyte count decreased (Investigations) | 2 (4)
Neutrophil count decreased (Investigations) | 3 (8)
Platelet count decreased (Investigations) | 3 (32)
White blood cell decreased (Investigations) | 3 (11)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (3)
Dizziness (Nervous system disorders) | 1 (2)
Paresthesia (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT03988205/Prot_SAP_000.pdf
  • Informed Consent Form: Subject Consent Form (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT03988205/ICF_001.pdf
  • Informed Consent Form: Caregiver Consent form (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT03988205/ICF_002.pdf